CLINICAL TRIAL: NCT00001582
Title: Collection of Blood, Bone Marrow and Tissue Samples for the Investigation of the Human Immune Response, Lymphoma Biology and HTLV-1 Infection
Brief Title: Investigation of the Human Immune Response in Normal Subjects and Patients With Disorders of the Immune System and Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970143; 97-C-0143; NCT00899067 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: T-cell Lymphoma; B-Cell Lymphoma; ATL; Myeloma
Keywords: Autoimmune Disorder; Immune System Evaluation; Human Response Investigation; Tissue Acquisition; Natural History
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, B-Cell; Neoplasms, Plasma Cell; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, tissue, bone marrow aspirate and biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Suspected or known disorder of the immune system or cancer; or, known or potential carrier of autoimmune disorder or immunodeficiency disease.

SUMMARY:
This protocol is being submitted to consolidate, update, and expand two previously approved protocols (77-C-0066 and 82-C-0044) into a single protocol. The purpose of this study is to examine the factors involved in the regulation of the immune system of healthy individuals and to define the abnormalities in this regulation that underlies the immunological disorders of patients with a variety of immunodeficiency and malignant disorders. The studies will include the ex vivo phenotypic and functional analysis of the network of cells involved in humoral and cellular immune responses, and in vivo testing for the capacity to make delayed-type hypersensitivity and humoral responses following immunization with a variety of antigens. Individuals to be studied will include patients with a variety of malignancies and patients with primary and secondary immunodeficiency disorders. Selected family members or family members known to be genetic carriers of certain immunodeficiency diseases as well as normal, unrelated individuals will also be studied. A small number of procedures will be used including analysis of blood obtained by phlebotomy, apheresis, skin testing and recall antigens and immunization to assess humoral immunity....

DETAILED DESCRIPTION:
Background:

* The evaluation of the cells of the immune system and HTLV-1 infection has been a central focus of the Metabolism Branch for the past 30 years.
* Blood obtained by apheresis or blood drawing, skin biopsies and other tissues will be evaluated for abnormalities related to immunity, HTLV-1 infection and the immune system.
* Advances in the characterization of acquired genetic changes in tumor samples has

led to insights for the development of targeted therapy of malignancy

Objectives:

* To characterize the molecular biology and immunological features as well as the clinical course of individuals with suspected or known disorders of the immune system or cancer
* To define the nature of the immunological, genetic and epigenetic abnormalities in the cells of patients with immunodeficiency diseases associated with infections and/or a high incidence of malignancy and in patients with cancer.
* To obtain whole blood, plasma and leukocytes, as well as skin, lymph node and bone marrow biopsies on patients with immunodeficiency or cancer to investigate the immune system.

Eligibility:

* Subjects with cancer.
* Subjects with immunodeficiency.
* Subjects with HTLV-1 infection.

Design:

-This is a natural history study that permits tissue acquisition for analysis of the immune system and HTLV-1 infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet at least one of these criteria:

Have suspected or known disorder of the immune system or cancer

Be a known or potential carrier of autoimmune disorder or immunodeficiency disease. Specific disorders may include but are not limited to:

* X-linked (severe combined immunodeficiency)
* Autosomal recessive SCID
* X-linked CD40 ligand deficiency
* Common variable immunodeficiency
* Ataxia-telangiectasia
* Wiskott Aldrich syndrome
* DiGeorge syndrome
* Infection with HTLV-1

Age greater than or equal to 18 years.

Participant must be able to understand and sign informed consent.

Participants who will undergo apheresis must have hematocrit greater than 28%, and platelet count greater than 50,000.

Subjects for whom apheresis is desired but whose counts are lower than those above must be evaluated and approved by a Department of Transfusion Medicine consult physician.

Weight greater than 25 kg is necessary for apheresis.

EXCLUSION CRITERIA:

Overall Exclusion Criteria:

Pregnant women will not be eligible for any aspect of this protocol.

Exclusion Criteria for Apheresis Alone:

Any diagnosed medical condition which may be worsened by the apheresis procedure. Specifically the participant should not have any of the following:

1. Congestive Heart Failure
2. History of angina
3. Severe hypotension (at the discretion of the participant's physician, the apheresis staff and the attending physician from the Department of Transfusion Medicine (DTM) per DTM Standard Operating Policies.)
4. Poorly controlled hypertension (average baseline blood pressure greater than 160/90)
5. History of a coagulation protein disorder.

Pediatric patients (less than 18 years) will not undergo apheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical patients/population with a suspected or known disorder of the immune system or cancer per the eligibility criteria.@@@
Sampling Method: Non-Probability Sample
Enrollment: 902 (Actual)
Dates: Start 1997-06-07 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Create Biobank | Ongoing
  No statistical endpoints are identified for this study; the purpose of the study is to acquire information regarding various immunodeficiency syndromes, HTLV-1 infection and malignancies. The data collected will not be combined for a summary report of the entire study; however, reports for specific disease entities may be published.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP. @@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. @@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.@@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1997-C-0143.html